CLINICAL TRIAL: NCT05610202
Title: Phase I Clinical Trial of Tolerability and Pharmacokinetics of TQB3702 Tablets in Hematologic Tumor Subjects
Brief Title: Tolerability and Pharmacokinetics Study of TQB3702 Tablets in Hematologic Tumor Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3702-I-01
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-04

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB3702 tablets (Experimental): TQB3702 tablets were administered orally, 28 days as a treatment cycle until the progressive diseases or the investigator judges that it is not suitable for subject to continue to take this medicine.
  Interventions: Drug: TQB3702 tablets

INTERVENTIONS:
Drug: TQB3702 tablets — TQB3702 tablets are selective BTK inhibitors.

SUMMARY:
This project is an open, dose escalation and expansion phase I clinical study. The first phase is a dose escalation study, and the second phase is a dose expansion study based on the Maximum tolerated dose (MTD) / Recommended Phase II Dose (RP2D) obtained in the first phase. The purpose is to evaluate the tolerability and preliminary efficacy of TQB3702 tablets in hematological tumor subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily joined the study, signed informed consent form, and with good compliance.
* ≥18 years old and ≤ 80 years old; Eastern Cooperative Oncology Group (ECOG) physical status: 0-2; at least 3 months expected survival period.
* Clearly diagnosed recurrent / refractory hematological tumors that meet the WHO definition;
* At least 1 measurable lesion for efficacy evaluation.
* The function of main organs is normal.
* Female patients of childbearing age should agree to use contraceptive measures during the study period and for at least 6 months after study is stopped; a negative serum pregnancy test within 7 days prior to study enrollment and must be non-lactating subjects; male patients should agree to use contraception during the study period and for at least 6 months after study is stopped.

Exclusion Criteria:

* Patients has had or is currently having other malignant tumors within 3 years. The following two conditions can be included in the group: other malignant tumors treated with a single operation to achieved 5 consecutive years of disease free survival (DFS)s. Cured cervical carcinoma in situ, non-melanoma skin cancer, nasopharyngeal carcinoma and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)].
* Subjects with central nervous system aggression (CNS);
* Received allogeneic hematopoietic stem cell transplantation (allo-HSCT) or had active graft-versus-host disease (GVHD) requiring immunosuppressive therapy within 12 months before the first dose;
* Multiple factors that affect the absorption of oral medications (e.g., inability to swallow, chronic diarrhea, and intestinal obstruction);
* Unrelieved toxicity of ≥CTC AE grade 1 due to any previous treatment, excluding alopecia and fatigue;
* Major surgical treatment, open biopsy, and significant traumatic injury were received within 28 days before the start of study treatment.
* The presence of active or uncontrolled primary autoimmune cytopenia, including autoimmune hemolytic anemia (AIHA) and primary immune thrombocytopenia (ITP);
* Patients with evidence or history of bleeding constitution; Or any bleeding event (such as gastrointestinal bleeding) greater than or equal to CTC AE level 3 within 4 weeks before the first medication;
* Subjects had an arteriovenous thrombosis event within 6 months.
* Subjects have history of psychotropic substance abuse and are unable to abstain or have mental disorders;
* Subjects with any severe and/or uncontrolled disease.
* Within 2 weeks before the first treatment, the subjects had received proprietary Chinese medicines with anti-tumor indications specified in the NMPA approved drug instructions;
* Uncontrolled pleural effusion, pericardial effusion, or ascites that still require repeated drainage (investigator judgment);
* Study treatment related: subjects received live or mRNA vaccines within 4 weeks before the first treatment or were scheduled to receive live or mRNA vaccines during the study;
* Participated in clinical trials of other antitumor drugs within 4 weeks before the first treatment;
* According to the investigator's judgment, there are concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or subjects who are considered unsuitable for enrollment for other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 104 weeks
  To evaluate the maximum tolerated dose of TQB3702 tablets in the treatment of relapsed/refractory hematologic tumors.
Dose limited toxicity (DLT) | Baseline up to 104 weeks
  To evaluate the dose-limiting toxic dose of TQB3702 tablets in the treatment of relapsed/refractory hematologic tumors.
Recommended Phase II Dose (RP2D) | Baseline up to 104 weeks
  To evaluate the phase II recommended dose of TQB3702 tablets in the treatment of relapsed/refractory hematological tumors.

SECONDARY OUTCOMES:
Time to Reach the Maximum Plasma Concentration (Tmax)-single dose | before administration, 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72hours after administration.
  Time to Reach the Maximum Plasma Concentration after single dose
Time to Reach the Maximum Plasma Concentration (Tmax)-multiple dose | before administration (-1~0h), 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24 hours after administration at Day 8/15/28 of Cycle1, Day 28 of Cycle 6; when withdrawn from the group due to disease progression or at the end of study treatment.
  Time to Reach the Maximum Plasma Concentration after multiple dose
Maximum plasma concentration (Cmax)-Single dose | before administration, 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72hours after administration.
  Cmax is the maximum plasma concentration of TQB3702 after single dose
Maximum plasma concentration (Cmax)-Multiple dose | before administration (-1~0h), 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24 hours after administration at Day 8/15/28 of Cycle1, Day 28 of Cycle 6; when withdrawn from the group due to disease progression or at the end of study treatment.
  Cmax is the maximum plasma concentration of TQB3702 after multiple dose
Elimination half-life (t1/2)-Single dose | before administration, 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72 hours after administration.
  t1/2 is time it takes for the blood concentration of TQB3702 or metabolite(s) to drop by half after single dose.
Elimination half-life (t1/2)-Multiple dose | before administration (-1~0h), 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24 hours after administration at Day 8/15/28 of Cycle1, Day 28 of Cycle 6; when withdrawn from the group due to disease progression or at the end of study treatment.
  t1/2 is time it takes for the blood concentration of TQB3702 or metabolite(s) to drop by half after multiple dose.
Area under the plasma concentration-time curve from time zero to time t (AUC0-t)-Single dose | before administration, 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72hours after administration.
  To characterize the pharmacokinetics of TQB3702 by assessment of area under the plasma concentration time curve from the first dose to a certain time.
Area under the plasma concentration-time curve from time zero to time t (AUC0-t)-Multiple dose | before administration (-1~0h), 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24 hours after administration at Day 8/15/28 of Cycle1, Day 28 of Cycle 6; when withdrawn from the group due to disease progression or at the end of study treatment.
  To characterize the pharmacokinetics of TQB3702 by assessment of area under the plasma concentration time curve from the first dose to a certain time.
Maximum (peak) steady-state plasma drug concentration during a dosage interval (Cmax,ss)-Single dose | before administration, 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72hours after administration.
  Maximum (peak) steady-state plasma drug concentration during a dosage interval (Cmax,ss) after Single dose
Maximum (peak) steady-state plasma drug concentration during a dosage interval (Cmax,ss)-Multiple dose | before administration (-1~0h), 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24 hours after administration at Day 8/15/28 of Cycle1, Day 28 of Cycle 6; when withdrawn from the group due to disease progression or at the end of study treatment.
  Maximum (peak) steady-state plasma drug concentration during a dosage interval (Cmax,ss) after Multiple dose
steady state area under the concentration-time curve over a dosing interval (AUCtau, ss)-single dose | before administration, 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72hours after administration.
  steady state area under the concentration-time curve over a dosing interval (AUCtau, ss) after single dose
steady state area under the concentration-time curve over a dosing interval (AUCtau, ss)-multiple dose | before administration (-1~0h), 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24 hours after administration at Day 8/15/28 of Cycle1, Day 28 of Cycle 6; when withdrawn from the group due to disease progression or at the end of study treatment.
  steady state area under the concentration-time curve over a dosing interval (AUCtau, ss) after multiple dose
Minimum steady-state plasma drug concentration during a dosage interval (Css-min)-Single dose | before administration, 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24, 48, 72hours after administration.
  Minimum steady-state plasma drug concentration during a dosage interval (Cmin-ss) after Single dose
Minimum steady-state plasma drug concentration during a dosage interval (Css-min)-multiple dose | before administration (-1~0h), 0.25, 0.5, 0.75, 1, 2, 4, 6, 12, 24 hours after administration at Day 8/15/28 of Cycle1, Day 28 of Cycle 6; when withdrawn from the group due to disease progression or at the end of study treatment.
  Minimum steady-state plasma drug concentration during a dosage interval (Cmin-ss) after multiple dose
Objective Response Rate (ORR) | Baseline up to 104 weeks
  The proportion of patients with tumor size reduction of a predefined amount and for a minimum time period
Complete Remission Rate (CRR) | Baseline up to 104 weeks
  The proportion of tumors that have a complete response after treatment
Disease Control Rate (DCR) | Baseline up to 104 weeks
  The percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease to a cancer treatment in clinical trials.
Duration of Response (DOR) | Baseline up to 104 weeks
  The time from the date of first documentation of a CR or PR or PD to the date of first documentation of tumor progression.
Progression Free Survival (PFS) | Baseline up to 104 weeks
  The time from the first dose to the first documentation of progressive disease (PD) or death from any cause, whichever occurs first
Overall Survival (OS) | Baseline up to 104 weeks
  the time from start of study treatment to date of death due to any cause
Adverse events (AE) | Baseline up to 104 weeks
  The occurrence of all adverse events (AE)
Serious adverse events (SAE) | Baseline up to 104 weeks
  The occurrence of all serious adverse events (SAE)
Bruton's tyrosine kinase (BTK) occupancy | Baseline up to 104 weeks
  The BTK occupancy in peripheral blood mononuclear cell (PMBC)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Cancer Hospital Affiliated to Shandong First Medical University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No